CLINICAL TRIAL: NCT00866125
Title: Hand Function, Health Related Quality of Life and Activity Performance in Patients With Polymyositis or Dermatomyositis.
Brief Title: Hand Function in Patients With Poly- or Dermatomyositis
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Ingrid Lundberg, Rheumatology unit, Department of Medicine.
Other Study IDs: 02-078
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: Polymyositis; Dermatomyositis; Grip force; Quality of life; Activity performance
MeSH Terms: conditions — Polymyositis; Dermatomyositis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate the hand function in patients with poly-and dermatomyositis and compare this to healthy individuals and norm values and secondly if hand function correlates to activity performance and health related quality of life.

The study is a cross-sectional study. To assess hand function the investigators will measure grip force with Grippit and arm/hand mobility using EPM-ROM scale. The activity performance will be measured with Myositis Activities Profile and health related quality of life will be assessed with SF-36.

The investigators' hypothesis is that hand function is reduced in comparison to the healthy population and that hand function affects both activity performance and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with definite or probable polymyositis or dermatomyositis (according to criteria by Bohan and Peter) were included in the study

Exclusion Criteria:

* Other diseases or injuries that could affect arm/hand mobility and grip force for example other rheumatological or neurological disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 patients diagnosed with polymyositis or dermatomyositis were identified through the myositis registry at the rheumatology clinic at Karolinska University Hospital, Stockholm, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2002-04; Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid E Lundberg, MD, PhD, Study Director — Karolinska Institutet